CLINICAL TRIAL: NCT05138341
Title: Hyperacute mEchAnicaL Endoscopic Minimally Invasive Surgical (MIS) Intracranial Hemorrhage Evacuation
Brief Title: Minimal Invasive Surgical Intracerebral Hemorrhage Removal
Acronym: HEALME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Dr. Richard Aviv, Head of Medical Imaging, The Ottawa Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210235-01H
Record Dates: First submitted 2021-10-12; First posted 2021-11-30 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Intracranial Hemorrhages
Keywords: Intracranial Hemorrhages; Minimally invasive hematoma evacuation; Hyperacute
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either minimally invasive hematoma evacuation with the Artemis Neuro Evacuation Device with medical management (MIS group) or best medical management alone (3:1) (MM)
Who Masked: Outcomes Assessor
Masking Description: D90 evaluations of mRS, NIHSS, Barthel Index will be performed by an evaluator blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Minimal Invasive Surgical (MIS) management (Experimental): Minimally invasive hematoma evacuation with the Artemis Neuro Evacuation Device with medical management
  Interventions: Device: Minimally invasive surgical (MIS) intracranial hemorrhage Evacuation
- Best Medical Management (MM) (No Intervention): Best medical management per standard of care

INTERVENTIONS:
Device: Minimally invasive surgical (MIS) intracranial hemorrhage Evacuation — Patients randomized to MIS group will be undergoing an intervention will get Minimal Invasive Surgical treatment.
  The market approved Artemis Device (MIS group) will be used. The Artemis Device, Aspiration Pump, and endoscope are used to rinse (irrigate) this area and to gently suction out the rinsing fluid and any blood or clot in brain. The Device is also designed to prevent clogging during the suction of fluid and blood.
  Arms: Mechanical Minimal Invasive Surgical (MIS) management

SUMMARY:
This is a feasibility study trial to determine whether hyperacute (≤8 hour) mechanical Minimal Invasive Surgical (MIS) management is feasible and secondarily improves outcome in patients with spontaneous supratentorial intracranial hemorrhage (ICH).

Patients meeting the inclusion and exclusion criteria, will be enrolled and randomized to either minimally invasive hematoma evacuation (MIS) or best medical management alone (MM). Subjects will be randomly assigned by a central web-based system in a 3:1 manner to treatment with MIS or MM. Data for each subject will be collected at the time of enrollment and treatment, and at subsequent follow-up visits.

DETAILED DESCRIPTION:
The proposed study seeks to determine whether hyperacute (≤8 hour) mechanical MIS management is feasible and improves outcome in patients with spontaneous supratentorial intracranial hemorrhage (ICH).

* Screening The subject will be evaluated as any non-traumatic spontaneous intra-parenchymal hemorrhage patient including medical history screened, available clinical/neurological exams (focused exam, NIHSS, GCS, historical mRS), ECG, laboratory work, and imaging information per institutional standard of care. A CTA (or MRA) will be performed, as standard of care.
* Randomization After all inclusion and exclusion criteria are confirmed and written informed consent obtained, randomization will occur. Subjects will be randomized to best MM or MIS.
* Treatment Procedure (if randomized to MIS) Minimally Invasive Surgical evacuation.
* Treatment Procedure (if randomized to MM) There is no intervention for the control group beyond the current standard of care provided at The Ottawa Hospital. Subjects randomized to the MM group will receive best MM for ICH according to Canadian Best Practice Recommendations for ICH care. Outcomes assessments will be in accordance to table 2.
* Post procedure, D1, D2 and D5 or discharging A post-procedural computed tomographic scan will be obtained within 24 hours (± 6 hours) for MIS group. Clinical assessment such as NIHSS, mRS, NCCT head, computed tomographic Angiogram, adverse event assessment will be conducted as SOC for MIS group (Table 2 in protocol).

A CT will be obtained in MM subjects 24 hours (± 6 hours) after randomization. Adverse event assessment will be conducted for MM subjects 4-6 hours after randomization. Neurological and functional exams will be conducted in D1 and D2 after randomization (Table 2 in protocol).

Follow-up visits (D30, D90): (Both MIS and MM groups) Follow-ups will be combined with phone and onsite visit. D30 will be conducted over the phone, and D90 will be onsite visit. The follow-ups will involve clinical assessment such as NIHSS, Glasgow Coma Scale, EuroQol- 5 Dimension (EQ-5D), mRS, Barthel, Glasgow Outcome Scale (GOSE), adverse event assessment, concomitant. medications.

ELIGIBILITY:
Inclusion Criteria:

1. CT diagnosed acute spontaneous primary supratentorial ICH.
2. Age >18 years
3. Baseline ICH volume 20-80 ml, estimated using the standard "A*B*C/2"calculation on the baseline CT.
4. NIHSS≥6 and Glasgow Coma Scale score 8-12, on initial screening.
5. Premorbid Modified Rankin score (MRS) ≤1
6. Systolic blood pressure140-180 millimeters of mercury (mmHg) with 160mmHg target according to practice guidelines
7. Randomize and first evacuation attempt ≤8 hours onset using the "last seen normal" principle.
8. Consent obtained from patient or their Substitute Decision Maker prior to enrolment.

Exclusion Criteria:

1. Infratentorial ICH (Brainstem or cerebellum).
2. ICH secondary to known or suspected trauma, aneurysm, vascular malformation, hemorrhagic conversion of ischemic stroke, venous sinus thrombosis, thrombolytic treatment, tumour, or infection; or an in-hospital ICH or ICH because of any in-hospital procedure or illness.
3. Baseline brain imaging shows evidence of acute or subacute ischemic stroke (chronic infarcts are not an exclusion).
4. Platelets <100000, International Normalized ratio (INR)>1.3 or clotting disorder. Coumadin reversal permitted if not required during hospitalization
5. Serious comorbidities including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, and hematologic disease or mechanical valve
6. Impaired brainstem function (bilateral fixed dilated pupils, extensor posturing).
7. Patient considered unstable in opinion of investigator.
8. Positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrolment <=8 hours | Baseline
  Number of patients eligible for treatment recruited
Number of patients with good functional outcome | Day 1 (baseline), Day 30 and Day 90
  Functional outcome assessed via modified Rankin score (mRS). Change from Day 1 to Day 90 will be assessed (0 no symptoms - 5 severe disability)
Quality of life assessment | Day 1, Day 5 and Day 90
  Quality of life assessed via NIH Stroke Scale 0: No stroke symptoms 1-4: Minor stroke 5-15: Moderate stroke 16-20: Moderate to severe stroke 21-42: Severe stroke Change from Day 1 to Day 90 will be assessed as well
Rate of mortality | Day 7
  Number of deaths
Rate of mortality | Day 30
  Number of deaths
Quality of life EQ-5D-5L | Day 90
  EQ-5D-5L stands for European Quality of Life Five Dimension, the 5-level EQ-5D version (EQ-5D-5L), which was introduced by European Quality of Life Scale group in 2009. EQ-5D-5L is used for self-assessment on activities of daily living.
  The EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels:
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems

SECONDARY OUTCOMES:
Cost-effectiveness analysis | Day 90
  Costs and outcomes will be assessed within 90 days to compare total costs and health outcomes of mechanical minimal Invasive Surgical Management and Best Medical Management.
Number of patients identifying deferred consent in ICH as acceptable | 1-2 years
  Investigators will secondarily explore the applicability, acceptability, and effects of implementing a deferral of consent policy in an emergency stroke trial.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aviv, MD, Principal Investigator — Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for primary and secondary outcomes will be made available.
Time Frame: The principal investigator will aim to have data available within 2 year of study completion
Access Criteria: Authors aim to have the study presented at conferences and published in a peer-reviewed journal.
  Participants can search this website to obtain study information.
URL: http://www.clinicaltrials.gov